CLINICAL TRIAL: NCT02799056
Title: Diaphragmatic Shortening Fraction and Pulmonary Ultrasound Combined Analysis for Extubation Success Prediction in Critical Care Patients
Brief Title: Diaphragmatic and Pulmonary US for Extubation Success Prediction
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Julio Edgardo González Aguirre, Dr., Hospital Universitario Dr. Jose E. Gonzalez
Other Study IDs: NM16-00003
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Airway Extubation
Keywords: Airway Extubation; Ultrasonography; Ventilator Weaning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Thoracic ultrasound — The ultrasound will be performed using the ultrasound system GE Logiq XP equipped with a linear probe of 10 MHz. The diaphragm is visualized as two parallel echogenic lines at the eighth intercostal space in the mid-axillary line. The images will be captured during the inspiratory and expiratory tidal volume to and during maximum inspiration and expiration. Each image will be frozen in B mode and the diaphragm thickness will be measured from the center line pleural half the peritoneal line. The fraction of diaphragmatic thickening it is calculated by the formula: diaphragmatic thickness at the end of inspiration - thickness to diaphragmatic at the end of exhalation / diaphragmatic thickness at the end of exhalation x 100. The number of areas with lines B also will be measured.

SUMMARY:
The primary objective is to assess whether the fraction of diaphragmatic shortening in combination with the presence / absence of alveolar-interstitial syndrome evaluated through chest ultrasound may predict successful extubation in adult patients hospitalized in the intensive care unit.

DETAILED DESCRIPTION:
The primary objective is to assess whether the fraction of diaphragmatic shortening in combination with the presence / absence of alveolar-interstitial syndrome evaluated through chest ultrasound may predict successful extubation in adult patients hospitalized in the intensive care unit. The investigators' null hypothesis is the fraction of diaphragmatic shortening in combination with the presence / absence of alveolar-interstitial syndrome evaluated through chest ultrasound can not predict the success of extubation in adult patients hospitalized in the intensive care unit.

The alternative hypothesis is the fraction of diaphragmatic shortening in combination with the presence / absence of alveolar-interstitial syndrome evaluated through chest ultrasound may predict successful extubation in adult patients hospitalized in the intensive care unit.

The study is a no experimental study of diagnostic test, prospective with longitudinal capture. The study will consist of two parts: the first with the aim of finding the values best combination of sensitivity and specificity compared to extubation success for diaphragmatic shortening fraction and the number of lung quadrants with lines B. In the second part the study will make the prospective validation of these values.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of older
* Hospitalized in medical or surgical intensive care unit
* Successful spontaneous ventilation trial

Exclusion Criteria:

* Patients reintubated after a first failure after extubation
* Injuries to prevent conduct ultrasound
* Pregnancy
* History of neuromuscular disease
* Brain injury that prevented adequate protection of the airway (Glasgow Coma Scale <8)
* Unilateral or bilateral Pneumothorax
* Presence of chest tube in right hemothorax
* Right subphrenic abscess
* Known uni- or bilateral phrenic nerve injury
* Unilateral or bilateral diaphragmatic Paralysis
* Unwillingness of the patient or guardian to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years or older patients, hospitalized in medical or surgical intensive care unit of the University Hospital "Dr. José E. González "from 1 may 2016 until the sample size is completed and who have successful spontaneous ventilation trial as part of routinely applied extubation protocol.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2016-05; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Extubation success | 72 h after extubation
  The investigators consider successful extubation when the patient does not require reintubation within 72 hours of its extubation

CONTACTS AND LOCATIONS:
Overall Officials: Julio E González, MD, Study Director — Universidad Autónoma de Nuevo León
Locations (1):
- UANL University Hospital, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] McConville JF, Kress JP. Weaning patients from the ventilator. N Engl J Med. 2012 Dec 6;367(23):2233-9. doi: 10.1056/NEJMra1203367. No abstract available. PMID 23215559
- [Background] Ely EW, Baker AM, Dunagan DP, Burke HL, Smith AC, Kelly PT, Johnson MM, Browder RW, Bowton DL, Haponik EF. Effect on the duration of mechanical ventilation of identifying patients capable of breathing spontaneously. N Engl J Med. 1996 Dec 19;335(25):1864-9. doi: 10.1056/NEJM199612193352502. PMID 8948561
- [Background] Yang KL, Tobin MJ. A prospective study of indexes predicting the outcome of trials of weaning from mechanical ventilation. N Engl J Med. 1991 May 23;324(21):1445-50. doi: 10.1056/NEJM199105233242101. PMID 2023603
- [Background] Huaringa AJ, Wang A, Haro MH, Leyva FJ. The weaning index as predictor of weaning success. J Intensive Care Med. 2013 Nov-Dec;28(6):369-74. doi: 10.1177/0885066612463681. Epub 2012 Oct 22. PMID 23753219
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Background] Lichtenstein DA, Meziere GA. Relevance of lung ultrasound in the diagnosis of acute respiratory failure: the BLUE protocol. Chest. 2008 Jul;134(1):117-25. doi: 10.1378/chest.07-2800. Epub 2008 Apr 10. PMID 18403664
- [Background] Silva S, Biendel C, Ruiz J, Olivier M, Bataille B, Geeraerts T, Mari A, Riu B, Fourcade O, Genestal M. Usefulness of cardiothoracic chest ultrasound in the management of acute respiratory failure in critical care practice. Chest. 2013 Sep;144(3):859-865. doi: 10.1378/chest.13-0167. PMID 23670087
- [Background] Enghard P, Rademacher S, Nee J, Hasper D, Engert U, Jorres A, Kruse JM. Simplified lung ultrasound protocol shows excellent prediction of extravascular lung water in ventilated intensive care patients. Crit Care. 2015 Feb 6;19(1):36. doi: 10.1186/s13054-015-0756-5. PMID 25656060
- [Background] Mongodi S, Via G, Bouhemad B, Storti E, Mojoli F, Braschi A. Usefulness of combined bedside lung ultrasound and echocardiography to assess weaning failure from mechanical ventilation: a suggestive case*. Crit Care Med. 2013 Aug;41(8):e182-5. doi: 10.1097/CCM.0b013e31828e928d. PMID 23863255
- [Background] Soummer A, Perbet S, Brisson H, Arbelot C, Constantin JM, Lu Q, Rouby JJ; Lung Ultrasound Study Group. Ultrasound assessment of lung aeration loss during a successful weaning trial predicts postextubation distress*. Crit Care Med. 2012 Jul;40(7):2064-72. doi: 10.1097/CCM.0b013e31824e68ae. PMID 22584759
- [Background] Jiang JR, Tsai TH, Jerng JS, Yu CJ, Wu HD, Yang PC. Ultrasonographic evaluation of liver/spleen movements and extubation outcome. Chest. 2004 Jul;126(1):179-85. doi: 10.1378/chest.126.1.179. PMID 15249460
- [Background] Boussuges A, Gole Y, Blanc P. Diaphragmatic motion studied by m-mode ultrasonography: methods, reproducibility, and normal values. Chest. 2009 Feb;135(2):391-400. doi: 10.1378/chest.08-1541. Epub 2008 Nov 18. PMID 19017880
- [Background] Ferrari G, De Filippi G, Elia F, Panero F, Volpicelli G, Apra F. Diaphragm ultrasound as a new index of discontinuation from mechanical ventilation. Crit Ultrasound J. 2014 Jun 7;6(1):8. doi: 10.1186/2036-7902-6-8. eCollection 2014. PMID 24949192
- [Background] Kim WY, Suh HJ, Hong SB, Koh Y, Lim CM. Diaphragm dysfunction assessed by ultrasonography: influence on weaning from mechanical ventilation. Crit Care Med. 2011 Dec;39(12):2627-30. doi: 10.1097/CCM.0b013e3182266408. PMID 21705883
- [Background] DiNino E, Gartman EJ, Sethi JM, McCool FD. Diaphragm ultrasound as a predictor of successful extubation from mechanical ventilation. Thorax. 2014 May;69(5):423-7. doi: 10.1136/thoraxjnl-2013-204111. Epub 2013 Dec 23. PMID 24365607
- [Background] Criner GJ. Measuring diaphragm shortening using ultrasonography to predict extubation success. Thorax. 2014 May;69(5):402-4. doi: 10.1136/thoraxjnl-2013-204920. No abstract available. PMID 24727579
- [Background] Diederich S, Link TM, Zuhlsdorf H, Steinmeyer E, Wormanns D, Heindel W. Pulmonary manifestations of Hodgkin's disease: radiographic and CT findings. Eur Radiol. 2001;11(11):2295-305. doi: 10.1007/s003300100866. PMID 11702175